CLINICAL TRIAL: NCT02622204
Title: The Effect of Corrective Osteotomy on in Vivo Cartilage Mechanobiology in Patients With Knee Osteoarthritis: Cross-sectional Observational Single-centre Study
Brief Title: The Effect of Corrective Osteotomy on in Vivo Cartilage Mechanobiology in Patients With Knee Osteoarthritis
Acronym: Osteotomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2015-224
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, synovium biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Corrective osteotomy: patients with knee osteoarthritis undergoing corrective osteotomy
  Interventions: Procedure: Corrective osteotomy

INTERVENTIONS:
Procedure: Corrective osteotomy — corrective osteotomy for varus alignment
  Other Names: Corrective osteotomy (CO)

SUMMARY:
Our overall hypothesis is that a sudden ambulatory load reduction (caused by corrective osteotomy) leads to changes in cartilage biology that delay or reverse osteoarthritic processes determining the clinical outcome and representing an in vivo model for assessing cartilage mechanosensitivity.

DETAILED DESCRIPTION:
Although osteoarthritis (OA) is the most common degenerative joint disease and despite international research efforts, to date the factors involved in the initiation and progression of this debilitating disease are poorly understood, diagnostic markers are lacking and there is no cure. High tibial osteotomy (HTO) is a well-accepted therapy for patients with knee OA and varus alignment aimed at re-establishing a more even distribution of ambulatory load between the affected medial knee compartment and the lateral knee compartment. However, the survival rate of HTO is only around 75% after 5 years. There is some evidence that the change in ambulatory load after HTO may be more relevant than the post-operative static alignment although this relationship has not yet been investigated. Because of the large changes in ambulatory load with HTO, the investigators propose that corrective osteotomy may serve as a valuable model for studying the effect of changes in ambulatory load on in vivo cartilage mechanobiology in patients with knee osteoarthritis. Our previous work has shown that serum biomarkers for cartilage increase after a 30-minute walking exercise (termed 'walking stress test') and indicated that these changes may be associated with the accumulated ambulatory load during the test.

Patients with medial compartment knee OA and varus alignment will be clinically assessed (including mechanical axis measurement from radiographs) and complete questionnaires on physical function prior to corrective osteotomy. Patients will complete a walking stress test with blood sampling to assess load-induced changes in serum biomarker concentrations, and undergo gait analysis to assess the external knee adduction moment. Once full load bearing is achieved, the mechanical axis will be measured from radiographs. Patients will complete the questionnaires and a second walking stress test with blood sampling and undergo gait analysis 6 months after corrective osteotomy. At the 12-month follow-up, subjects will complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* radiographically diagnosed and isolated symptomatic medial compartment knee OA undergoing corrective osteotomy (Kellgren-Lawrence grade 2 or 3)
* pain level not limiting physical activity participation
* sports participation (at least once/week).

Exclusion Criteria:

* Use of walking aids
* inability to walk for 30 minutes
* age < 18 years (before maturation) or age >70 years
* due to advanced general sarcopenia (degenerative loss of muscle mass in aging)
* body mass index (BMI) > 35 kg/m2
* active rheumatic disorder
* prior neuromuscular impairment (e.g. stroke)
* conditions other than knee OA that could cause abnormal patterns of locomotion
* prior hip, knee, and ankle prosthesis or osteotomy of the lower extremities
* prior spine surgery; other major medical problems
* investigators and their immediate families are not permitted to be subjects
* persons who have previously completed or withdrawn from this study
* patients currently enrolled in another experimental (interventional) protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with knee osteoarthritis scheduled for corrective osteotomy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change in load-induced biomarker concentration | 6 months

SECONDARY OUTCOMES:
knee adduction moment | 6 months
  knee adduction moment during walking
mechanical axis alignment | 6 months
knee osteoarthritis outcome scale | 12 months
synovial fluid biomarker concentration | 0 months
level of synovial inflammation | 0 months
level of gene expression | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinic for Orthopaedics and Traumatology, University Hospital basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mundermann A, Nuesch C, Herger S, Liphardt AM, Chammartin F, De Pieri E, Egloff C. Load-induced blood marker kinetics in patients with medial knee compartment osteoarthritis are associated with accumulated load and patient reported outcome measures. F1000Res. 2024 Jan 12;12:299. doi: 10.12688/f1000research.131702.2. eCollection 2023. PMID 38882712
- [Derived] De Pieri E, Nuesch C, Pagenstert G, Viehweger E, Egloff C, Mundermann A. High tibial osteotomy effectively redistributes compressive knee loads during walking. J Orthop Res. 2023 Mar;41(3):591-600. doi: 10.1002/jor.25403. Epub 2022 Jul 6. PMID 35730475